CLINICAL TRIAL: NCT01774474
Title: PRevention of Macular EDema After Cataract Surgery
Acronym: PREMED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: European Society of Cataract and Refractive Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NL42463.068.12
Record Dates: First submitted 2013-01-07; First posted 2013-01-24 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2016-05

CONDITIONS: Cystoid Macular Edema; Cataract; Diabetes Mellitus
Keywords: Prevention
MeSH Terms: conditions — Macular Edema; Cataract; Diabetes Mellitus | interventions — bromfenac; Dexamethasone; Bevacizumab; Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Non diabetics: bromfenac (Active Comparator): bromfenac 0.09% eye drops twice daily starting two days before surgery and continuing 2 weeks postoperatively
  Interventions: Drug: Bromfenac
- Non diabetics: dexamethasone (Active Comparator): dexamethasone 0.1% eye drops four times daily starting two days before surgery and continuing four times daily during the first postoperative week and one drop less per day every following week
  Interventions: Drug: Dexamethasone
- Non diabetics: bromfenac & dexamethasone (Active Comparator): bromfenac 0.09% eye drops twice daily starting two days before surgery and continuing 2 weeks postoperative & dexamethasone 0.1% eye drops four times daily starting two days before surgery and continuing four times daily during the first postoperative week and one drop less per day every following week
  Interventions: Drug: Bromfenac; Drug: Dexamethasone
- Diabetics: eye drops (Active Comparator): bromfenac 0.09% eye drops twice daily starting two days before surgery and continuing 2 weeks postoperative & dexamethasone 0.1% eye drops four times daily starting two days before surgery and continuing four times daily during the first postoperative week and one drop less per day every following week
  Interventions: Drug: Bromfenac; Drug: Dexamethasone
- Diabetics: eye drops & TA (Active Comparator): bromfenac 0.09% eye drops twice daily starting two days before surgery and continuing 2 weeks postoperative & dexamethasone 0.1% eye drops four times daily starting two days before surgery and continuing four times daily during the first postoperative week and one drop less per day every following week
  & a peroperative subconjunctival injection of 40 mg triamcinolone acetonide (TA, Triesence/Vistrec)
  Interventions: Drug: Bromfenac; Drug: Dexamethasone; Drug: Triamcinolone Acetonide
- Diabetics: eye drops & bevacizumab (Active Comparator): bromfenac 0.09% eye drops twice daily starting two days before surgery and continuing 2 weeks postoperative & dexamethasone 0.1% eye drops four times daily starting two days before surgery and continuing four times daily during the first postoperative week and one drop less per day every following week
  & a peroperative intravitreal injection of 1.25 mg bevacizumab (Avastin)
  Interventions: Drug: Bromfenac; Drug: Dexamethasone; Drug: Bevacizumab
- Diabetics: eye drops, TA & bevacizumab (Active Comparator): bromfenac 0.09% eye drops twice daily starting two days before surgery and continuing 2 weeks postoperative, dexamethasone 0.1% eye drops four times daily starting two days before surgery and continuing four times daily during the first postoperative week and one drop less per day every following week
  & a peroperative subconjunctival injection of 40 mg triamcinolone acetonide (TA)
  & a peroperative intravitreal injection of 1.25 mg bevacizumab
  Interventions: Drug: Bromfenac; Drug: Dexamethasone; Drug: Bevacizumab; Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Bromfenac
  Other Names: Yellox; Product code: EMEA/H/C/001198
  Arms: Diabetics: eye drops; Diabetics: eye drops & TA; Diabetics: eye drops & bevacizumab; Diabetics: eye drops, TA & bevacizumab; Non diabetics: bromfenac; Non diabetics: bromfenac & dexamethasone
Drug: Dexamethasone
  Other Names: Dexamethasone ophthalmic solution; Product code (NL): RVG 56003
  Arms: Diabetics: eye drops; Diabetics: eye drops & TA; Diabetics: eye drops & bevacizumab; Diabetics: eye drops, TA & bevacizumab; Non diabetics: bromfenac & dexamethasone; Non diabetics: dexamethasone
Drug: Bevacizumab
  Other Names: Avastin; Product code: EU/1/04/300/002
  Arms: Diabetics: eye drops & bevacizumab; Diabetics: eye drops, TA & bevacizumab
Drug: Triamcinolone Acetonide
  Other Names: Triesence or Vistrec; Product code (NL): RVG 106092
  Arms: Diabetics: eye drops & TA; Diabetics: eye drops, TA & bevacizumab

SUMMARY:
Cystoid macular edema (CME) is a common cause of vision loss after cataract surgery. In the last few years, several new treatments have been tried to address the problem of CME after cataract surgery in diabetic and non-diabetic patients. The investigators will perform a large RCT with the aim to provide more definite evidence-based recommendations for clinical guidelines to prevent the occurrence of CME after cataract surgery in patients with and without diabetes mellitus (DM).

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effect of different preventive strategies on the occurrence of CME after cataract surgery in non-diabetic and diabetic patients. The design of the study is a multicentre randomised controlled clinical trial. The study population will consist of 926 non-diabetic patients and 209 patients with diabetes mellitus (DM) who require cataract surgery in at least one eye. All patients will receive a phacoemulsification for cataract and placement of a posterior chamber intraocular lens (IOL).

In the non-diabetic population, the patients will receive either bromfenac 0.09% eye drops twice daily starting two days before surgery and continuing 2 weeks postoperative, dexamethasone 0.1% eye drops four times daily starting two days before surgery and continuing four times daily during the first postoperative week and one drop less per day every following week or a combination of both drugs.

In the diabetic population patients will receive either:

* Topical bromfenac 0.09% and dexamethasone 0.1% in the aforementioned dose;
* Topical bromfenac 0.09% and dexamethasone 0.1% in the aforementioned dose and a subconjunctival injection of 40 mg triamcinolone acetonide;
* Topical bromfenac 0.09% and dexamethasone 0.1% in the aforementioned dose and an intravitreal injection of 1.25 mg bevacizumab;
* Topical bromfenac 0.09% and dexamethasone 0.1% in the aforementioned dose, a subconjunctival injection of 40 mg triamcinolone acetonide and an intravitreal injection of 1.25 mg bevacizumab.

The primary endpoint is the change in central subfield mean macular thickness in the 1 mm area (central subfield macular thickness, CSMT) as compared to baseline within the first 6 weeks postoperative.

The secondary endpoint is the occurrence of postoperative clinically significant macular edema (CSME) within 12 weeks postoperatively. Other study endpoints are mean CDVA in logMAR at 6 weeks and 12 weeks postoperatively; OCT measured average retinal thickness in the central inner circle (3mm), the outer circle (6mm), and the macular volume at 6 weeks and 12 weeks postoperatively; intraocular pressure at 6 weeks and 12 weeks postoperatively.

In case of clinically significant macular edema, treatment will be initiated and its effect will be part of the evaluation at 12 weeks. Medical data of all patients who develop macular edema during this study will be checked at least 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing routine phacoemulsification (one eye per patient)
* willing and/or able to comply with the scheduled visits and other study procedures.
* able to communicate properly and understand instructions.
* accepting possible off-label use of intravitreal bevacizumab and/or subconjunctival preservative-free TA.

Exclusion criteria will be different for non-diabetic and diabetic patients. All ophthalmic exclusion criteria are applicable to the study eye only, unless stated otherwise.

General exclusion criteria for participation in this study are:

1. age below 21 years old;
2. participation in another clinical study;
3. post-traumatic cataract;
4. combined surgery;
5. functional monoculus;
6. previous ocular surgery;
7. progressive glaucoma with severe visual field defects, use of anti-glaucomatous medication or steroid-induced IOP elevation that required IOP-lowering treatment;
8. IOP ≥ 25 mmHg;
9. history of any intraocular inflammation or uveitis;
10. history of pseudoexfoliation syndrome, which is expected to cause peroperative complications;
11. history of Fuchs' endothelial dystrophy or cornea guttata 3+;
12. history of retinal vein occlusion;
13. any macular pathology that might influence VA, other than DME;
14. use of intravitreal bevacizumab or ranibizumab in the previous 6 weeks or intravitreal aflibercept in the previous 10 weeks;
15. use of intra- or periocular corticosteroid injection in the previous 4 months;
16. current use of topical NSAIDs or corticosteroids;
17. use of systemic corticosteroids (≥ 20 mg prednisolone or equivalence);
18. history of relevant adverse events, including serious adverse events (SAE), occurring after administration of NSAIDs, acetylsalicylic acid, sodium sulphite, corticosteroids or bevacizumab;
19. contraindications for use of topical NSAIDs, topical or subconjunctival corticosteroids or intravitreal bevacizumab or related drugs;

Non-diabetic patients with a history of CME will be excluded from participation in the study.

Additionally, diabetic patients will be excluded from participation in case of:

1. macular edema with a CSMT ≥450 µm;
2. very severe NPDR or proliferative DR requiring panretinal photocoagulation or vitrectomy;
3. vitreous haemorrhage present during preoperative visit(s);
4. cerebrovascular accident (CVA), myocardial infarction (MI) or other thromboembolic events in the previous 3 months;
5. a history of recurrent thromboembolic events;
6. a history of severe systemic bleeding in the previous 3 months;
7. major surgery in the previous 3 months;
8. history of glaucoma;

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1127 (Actual)
Dates: Start 2013-07-10 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2016-11-04 (Actual)

PRIMARY OUTCOMES:
Change in central subfield mean macular thickness as a measurement of efficacy | 6 weeks postoperatively
  The primary endpoint is the change in central subfield mean macular thickness in the 1 mm area (central subfield macular thickness, CSMT) as compared to baseline within the first 6 weeks postoperatively.

SECONDARY OUTCOMES:
No. of subjects developing clinically significant macular edema as a measurement of efficacy | 12 weeks postoperatively
  The secondary endpoint is the occurrence of postoperative clinically significant macular edema (CSME) within 12 weeks postoperatively.

OTHER OUTCOMES:
Change in corrected distance visual acuity (CDVA) as a measurement of efficacy | 6 postoperatively
  CDVA measurements will be taken using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts (logMAR).
Change in retinal thickness in the central inner circle (3mm) as a measurement of efficacy | 6 weeks postoperatively
  Measured using Optical Coherence Tomography (OCT)
Intraocular pressure (IOP) as a measurement of safety | 6 postoperatively
  IOP (in mmHg) will be measured by Goldmann applanation tonometry
Health-related quality of life as a measurement of efficacy and tolerability | 12 weeks postoperatively
  Using the Health Utility Index mark 3 (HUI-3)
No. of subjects with Adverse Events as a measurement of safety and tolerability | 6 weeks postoperatively
  An adverse event (AE) is defined as any undesirable experience occurring to a subject during the study, whether or not considered related to the investigational product. All adverse events reported spontaneously by the subject or observed by the principal investigator or his staff will be recorded.
  Most frequently reported adverse events which might occur while using the study medication: abnormal sensation in the eye, pain or irritation, redness or headache while using eye drops; increased IOP and masking of infections while using corticosteroids; retinal detachment, thrombo-embolic events, endophthalmitis and anterior chamber reactions after intravitreal injections of bevacizumab.
Change in retinal thickness in the central outer circle (6mm) as a measurement of efficacy | 6 weeks postoperatively
  Using OCT
Change in macular volume as a measurement of efficacy | 6 postoperatively
  Using OCT
Vision-related quality of life as a measurement of efficacy and tolerability | 12 weeks postoperatively
  Using the National Eye Institute Visual Functioning Questionnaire 25 (NEI-VFQ 25)
Cost-effectiveness | 12 weeks postoperatively
  Incremental cost-effectiveness ratios of the costs per quality-adjusted life year (QALY) and costs per improved patient on the NEI VFQ-25 and HUI-3.
Change in corrected distance visual acuity (CDVA) as a measurement of efficacy | 12 weeks postoperatively
  CDVA measurements will be taken using ETDRS visual acuity testing charts (logMAR).
Change in retinal thickness in the central inner circle (3mm) as a measurement of efficacy | 12 weeks postoperatively
  Measured using Optical Coherence Tomography (OCT)
Intraocular pressure (IOP) as a measurement of safety | 12 weeks postoperatively
  IOP (in mmHg) will be measured by Goldmann applanation tonometry
No. of subjects with Adverse Events as a measurement of safety and tolerability | 12 weeks postoperatively
  An adverse event (AE) is defined as any undesirable experience occurring to a subject during the study, whether or not considered related to the investigational product. All adverse events reported spontaneously by the subject or observed by the principal investigator or his staff will be recorded.
  Most frequently reported adverse events which might occur while using the study medication: abnormal sensation in the eye, pain or irritation, redness or headache while using eye drops; increased IOP and masking of infections while using corticosteroids; retinal detachment, thrombo-embolic events, endophthalmitis and anterior chamber reactions after intravitreal injections of bevacizumab.
Change in retinal thickness in the central outer circle (6mm) as a measurement of efficacy | 12 weeks postoperatively
  Using OCT
Change in macular volume as a measurement of efficacy | 12 weeks postoperatively
  Using OCT
Change in central subfield mean macular thickness as a measurement of efficacy | 12 weeks postoperatively
  Using OCT

CONTACTS AND LOCATIONS:
Overall Officials: prof. Rudy MM Nuijts, MD, PhD, Principal Investigator — University Eye Clinic Maastricht, University Hospital Maastricht
Locations (16):
- Austria (2):
  - Vienna Institute for Research in Ocular Surgery, Hanusch Krankenhaus, Vienna
  - Hospital of the Brothers of Saint John of God, Vienna
- University Hospital Antwerp, Edegem, Belgium
- Goethe University, Frankfurt am Main, Germany
- Semmelweis University, Budapest, Hungary
- Netherlands (9):
  - VU University Medical Center, Amsterdam
  - Academic Medical Center, Amsterdam
  - Amphia Hospital Breda, Breda
  - Zuyderland Medical Center, Heerlen
  - Eye Hospital Zonnestraal, Hilversum
  - University Eye Clinic Maastricht UMC+, Maastricht
  - Medical Centre Haaglanden, The Hague
  - St. Elisabeth Hospital, Tilburg
  - Máxima Medical Center Veldhoven, Veldhoven
- University Hospital Coimbra, Coimbra, Portugal
- Instituto Microcirurgia Ocular, Barcelona, Spain

REFERENCES:
- [Derived] Simons RWP, Wielders LHP, Nuijts RMMA, Veldhuizen CA, van den Biggelaar FJHM, Winkens B, Schouten JSAG, Dirksen CD; ESCRS PREMED Study Group. Economic evaluation of prevention of cystoid macular edema after cataract surgery in diabetic patients: ESCRS PREMED study report 6. J Cataract Refract Surg. 2022 May 1;48(5):555-563. doi: 10.1097/j.jcrs.0000000000000785. PMID 34417781
- [Derived] Simons RWP, Wielders LHP, Dirksen CD, Veldhuizen CA, van den Biggelaar FJHM, Winkens B, Schouten JSAG, Nuijts RMMA; ESCRS PREMED Study Group. Economic evaluation of prevention of cystoid macular edema after cataract surgery in patients without diabetes: ESCRS PREMED study report 4. J Cataract Refract Surg. 2021 Mar 1;47(3):331-339. doi: 10.1097/j.jcrs.0000000000000449. PMID 33009281